CLINICAL TRIAL: NCT05221554
Title: Pre-Op Total Hip Arthroplasty Modelling: Individualized Care, Improved Outcomes
Brief Title: Pre-Op THA Modelling
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Brent Lanting, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11307
Record Dates: First submitted 2021-10-27; First posted 2022-02-03 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Total Hip Arthroplasty; Computer-Assisted Surgery
Keywords: Osteoarthritis; Joint Disease; Musculoskeletal Disease
MeSH Terms: conditions — Osteoarthritis; Joint Diseases; Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prospective Computer-Navigated Cohort (Experimental): Patients in this arm will receive standard patient of care implants but navigation software will be used to plan optimal acetabular cup placement.
  Interventions: Procedure: Computer-navigated THA surgery
- Cross-sectional Standard of Care Cohort (Active Comparator): Patients in this arm will receive standard of care implants and undergo standard of care procedure for total hip arthroplasty.
  Interventions: Procedure: Standard of care THA surgery

INTERVENTIONS:
Procedure: Computer-navigated THA surgery — Navigation software coupled with real-time modeling software will be used to plan optimal acetabular cup for patients undergoing THA.
  Arms: Prospective Computer-Navigated Cohort
Procedure: Standard of care THA surgery — Patients already underwent THA procedure with manual placement of acetabular cup with conventional instrumentation.
  Arms: Cross-sectional Standard of Care Cohort

SUMMARY:
Replacing diseased hip joints with prosthetic implants in a procedure called total hip arthroplasty (THA) is associated with high rates of patient satisfaction, pain relief, and functional improvement when the implant is appropriately placed. Incorrect implant size or placement may lead to a breadth of negative outcomes, which could result in the need for implant revision. It is difficult to assess the precise orientation of patient hips on the operating table, with one study revealing that only 26% of acetabular cups placed without technological assistance are correctly positioned. Using computer navigation as a guide to achieve optimal implant alignment may improve successful placement rates. The additional incorporation of real-time modeling software may further help realize higher rates of successful implant placement. This study, therefore, aims to investigate a computer navigation system coupled with real-time modeling software to establish the benefit of such technology in the operating room, and further improve positive patient outcomes following THA. We hypothesize that including technological assistance in THAs will yield better patient outcomes compared to surgeries performed freehand.

ELIGIBILITY:
Inclusion Criteria:

* osteoarthritis of the hip requiring primary THA
* 40 years of age or older
* BMI <40 kg/m2
* able to provide informed consent, able and willing to do study assessments and follow instructions

Exclusion Criteria:

* prior surgery on the indicated hip with insertion of hardware
* prior surgery on the lower spine with insertion of hardware
* hip and/or spinal fixed deformities or inflammatory/ossification processes of the spine (e.g. DISH, ankylosing spondylolisthesis)
* limitations to range of motion of the contralateral hip

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Acetabular cup position | 6 months post-op
  CT examination. Measuring acetabular cup inclination and anteversion in degrees.
Protrusion length | 6 months post-op
  CT examination. Length of protrusion in the sagittal and axial view.
Acetabular cup loosening | 6 months post-op
  CT examination. Presence od acetabular cup loosening, indicated by periprosthetic radiolucency > 2 mm in width.
Degree of heterotopic ossification | 6 months post-op
  CT examination. Classification of heterotopic ossification based on Brooker Classification.
Muscle area | 6 months post-op
  CT examination measuring muscle cross-sectional area (in mm2).
Muscle density | 6 months post-op
  CT examination measuring radiological density (in HU).
Capsular scarring | 6 months post-op
  MRI examination. Measuring the joint capsule in its thickest part.
Joint effusion. | 6 months post-op
  MRI examination. Grading according to Mitchel et al. 1986
Quantification of fluid. | 6 months post-op
  MRI examination. Grading according to Mitchel et al. 1986
Heterotopic ossification in periarticular soft tissues. | 6 months post-op
  MRI examination. Classification of heterotopic ossification based on Brooker Classification.
Soft tissue impingement | 6 months post-op
  MRI examination. Measuring acetabular angle of anteversion.
Integrity of the periarticular muscles. | 6 months post-op
  MRI examination. Grading based on the Goutallier classification.

SECONDARY OUTCOMES:
Oxford Hip Score | 3- and 6-months post-op
  Joint-specific patient-reported outcome measure of disability in patients following THA
UCLA Activity Score | 3- and 6-months post-op
  Validated 10-point scale evaluating patient activity levels
VR-12 | 3- and 6-months post-op
  Patient-reported outcome measure of patient's overall perspective of their health
WOMAC questionnaire | 3- and 6-months post-op
  Self-administered questionnaire assessing activities of daily living, functional mobility, gait, general health and quality of life.
Novel questionnaire | 3- and 6-months post-op
  Self-reported outcome measure that assess the patient's ability to perform 10 common activities of daily living (gait, pivot left, pivot right, upstairs, downstairs, step over, chair sit/rise, bend forward, sit low, and squat)
Harris Hip Score | 3- and 6-months post-op
  A measure of dysfunction following total hip arthroplasty

CONTACTS AND LOCATIONS:
Overall Officials: Brent Lanting, Principal Investigator — London Health Sciences Centre/Lawson
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No